CLINICAL TRIAL: NCT06053918
Title: Psychological Follow-up in a Protected Hematology Unit as a Transitional Device Between Hospitalization and Return Home
Brief Title: Research-Action in Hematology From Hospitalization to Home
Acronym: RAH HD
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 18-199
Record Dates: First submitted 2023-07-28; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-07

CONDITIONS: Hematologic Cancer
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- classic follow-up (Group A): Group A will benefit from the classic follow-up, as it has been contractualized for several years now between the UMDSP and the hematology sector. Namely a psychological follow-up in the patient's room during the hospitalization time, once a week, more if the patient is going through a difficult passage that requires closer support. This follow-up is spread over an approximate period of 6 weeks maximum, depending on the length of hospitalization
- Intervention group (Group B): Group B will benefit from this same follow-up, to which will be added an interview when leaving the sector, and the extension of follow-up of the patient at home according to the same conditions: once a week, more if necessary, over a period of two months. This follow-up is spread over an approximate period of 15 weeks maximum, depending on the length of hospitalization.
  Interventions: Other: additional follow-up extension at home

INTERVENTIONS:
Other: additional follow-up extension at home — additional interview when leaving the sector, and the extension of follow-up of the patient at home
  Groups: Intervention group (Group B)

SUMMARY:
Objective :

To study and support the hospitalization and the return home of patients with the help of a psychological follow-up started in a hospital institution and which will continue in the patient's home, based on the concepts of transitionality and narrativity.

Material and method To do this, the subjects will benefit from psychological interviews where they will freely discuss what concerns them, whether it is illness, treatment, returning home, or any other personal subject.

They will be divided into two groups of 5 patients each, one of the groups will benefit from follow-up in an institution as contracted for several years between the Institute of Hematology and the psychologists of the UMDSP, another from the same follow-up but with the presence of the psychologist at the time of discharge extended to the patient's home after leaving the hospital for a period of 2 months.

To ensure a certain consistency in the evaluation criteria, these will be standardized in the form of questionnaires completed blindly by the patient, a caregiver and the investigator, at 3 key times of the research (entry, discharge from hospital, two months after this discharge)

Device tested:

The aim of this work is to test the benefits of a device based on transitionality, which can limit, thanks to the restoration of the symbolization process, the deleterious effects of each of the stages imposed by the disease, the care and the resumption of autonomy once the active phase of care has passed.

Narrativity is also at the heart of this transitional device. It makes it possible to evoke the present experience of the patient in connection with future projects and in the continuity of past, potentially traumatic events. It opens onto a dynamic temporal perspective where the trauma freezes.

The whole process promotes the subjective reappropriation of the experience and a psychic well-being.

ELIGIBILITY:
Inclusion Criteria:

* patient hospitalized Protected Hematology Unit
* patient with haematologic cancer
* patient requesting psychological assistance or accepting proposed psychological assistance
* signed informed consent

Exclusion Criteria:

* patient refusing to participate
* patient not able to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patient in Protected Hematology Unit
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of the psychological state, anxiety-depressive disorders | At hospital Month 0 and at home Month 2
  anxiety-depressive disorders yes or no

CONTACTS AND LOCATIONS:
Locations (1):
- CAEN University Hospital, Caen, France